CLINICAL TRIAL: NCT01294202
Title: An Open-Label, Randomised, Multi-Centre, Phase II Study to Investigate the Safety and Efficacy of AT13387, Either as Monotherapy or in Combination With Imatinib, in Patients With Unresectable and/or Metastatic Malignant GIST Whose Tumour Has Progressed Following Treatment With a Maximum of Three Tyrosine Kinase Inhibitors
Brief Title: A Study to Investigate the Safety and Efficacy of AT13387, Alone or in Combination With Imatinib, in Patients With GIST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT13387/0002
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Gastrointestinal Stromal Tumor (GIST)
Keywords: GIST; Gastrointestinal Stromal Tumor; unresectable; metastatic; AT13387; Astex; Gleevec; Imatinib
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Neoplasm Metastasis | interventions — (2,4-dihydroxy-5-isopropylphenyl)-(5-(4-methylpiperazin-1-ylmethyl)-1,3-dihydroisoindol-2-yl)methanone; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AT13387 and imatinib (Experimental): AT13387 administered on days 1, 8 and 15, imatinib administered daily
  Interventions: Drug: AT13387 and Imatinib

INTERVENTIONS:
Drug: AT13387 and Imatinib — In part 1 pts will receive AT13387 in combination with imatinib. Up to 5 possible dose levels of AT13387 could be evaluated in combination with imatinib 400 mg daily: 120 mg/m2, 150 mg/m2, 180 mg/m2, 220 mg/m2 and 260 mg/m2. AT13387 IV (in the vein) on day 1, 8 and 15 of each 28 day cycle, until progression or unacceptable toxicity develops, in order to establish the recommended phase II combination dose, which will be used in part 2 and/or part 3 of the study.
  In part 2 an additional 6-9pts will be treated.
  In part 3, provided that sufficient evidence of anti-tumour effect was observed in part 2 (disease stabilisation or reduction in tumour dimensions by RECIST), then an additional 12pts will be treated with AT13387 in combination with imatinib. Alternatively, if combination treatment is found to have excellent efficacy the randomised phase of the study may start so that 12 pts receive AT13387 on its own (monotherapy) and 12 pts receive AT13387 in combination with imatinib.
  Other Names: Gleevec

SUMMARY:
The purpose of this study is to investigate if an investigational drug called AT13387 is active against Gastrointestinal Stromal Tumor (GIST) that is resistant to other treatments, and to understand more about the safety of AT13387.

Most subjects in the study will receive AT13387 along with another drug called imatinib (Gleevec). Imatinib is a standard (approved) drug for treating patients with GIST. Some patients may receive AT13387 on its own. As a result, we shall begin to understand the effects of AT13387 given on its own and when combined with imatinib.We shall also find out more about the side-effects of AT13387, and more about how the body breaks down (metabolizes) AT13387.

DETAILED DESCRIPTION:
The study consists of 3 parts: Part 1 is a dose escalation phase, Part 2 is a dose expansion phase and Part 3 is either a further dose expansion phase or a randomised phase in which half the patients receive AT13387 monotherapy and half continue to receive AT13387 in combination with imatinib.

All patients will receive AT13387 given by intravenous infusion on Days 1, 8, and 15 of a 28-day cycle. Most patients will also receive imatinib 400 mg by mouth every day.

Patients will have tumour imaging at baseline, and at 2, 4 and 6 months, and then at 2 month intervals until cycle 12, and then 3-monthly thereafter.

Blood samples will be taken to measure plasma drug levels of AT13387 given in combination with imatinib

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the risks of the study and to provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local subject privacy regulations).
* Age 18 years or older.
* Unresectable and/or metastatic malignant GIST with objective progression of disease following treatment with a maximum of 3 tyrosine kinase inhibitors (TKIs) including imatinib. To clarify, it is the number of TKIs - up to a maximum of three agents, including imatinib - that is the criterion for entry, not the number of prior courses of TKI treatment.
* Measurable disease.
* ECOG performance status 0 or 1.
* Negative blood or urine pregnancy test (within 7 days prior to commencing treatment), or documented evidence of surgical sterility, or natural or treatment-induced post-menopausal status with last menses >1 year ago.
* Willing to provide a tissue block or unstained slides of archived tumour for central pathology review and genotyping, or a full pathology report and results of genotyping of a previous tumour sample, or willing to undergo a new tumour biopsy for central pathology review and genotyping during the screening period of the study (prior to dosing)

Exclusion Criteria:

* Pregnancy or lactation (women of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to commencing treatment ). Male and female patients of childbearing potential must use appropriate birth control (abstinence, barrier methods, oral contraceptives and/or intrauterine devices) during the entire duration of the study, or the patient must be surgically sterile (with documentation in the patient's medical records).
* Impaired liver function, as evidenced by prior liver segmentectomy or hemi-hepatectomy; or alanine or aspartate aminotransferase (ALAT/ASAT) >2.5x ULN; or alkaline phosphatase >2.0x ULN; or bilirubin >2.0x ULN.
* Abnormal clotting, as evidenced by PT or PTT >1.5x ULN, or therapeutic/prophylactic anticoagulation.
* Renal impairment, defined as either serum creatinine higher than the institution ULN,or estimated creatinine clearance lower than LLN (i.e. patients should have both normal serum creatinine, and normal estimated creatinine clearance)
* Impaired marrow function, defined as haemoglobin <9.0 g/dL, neutrophils <1.5 x10^9/L, or platelets <100 x10^9/L. Patients may receive a blood transfusion for anaemia to allow entry to the study but should not be transfusion-dependent.
* Left ventricular ejection fraction <50% on echocardiography or MUGA scan.
* Known metastases of the central nervous system.
* Prior anticancer therapies including tyrosine kinase inhibitors (other than imatinib) not completed within 2 weeks or 5 half-lives of the agent (including known active metabolites) prior to treatment with study drug. Patients receiving imatinib should continue to receive imatinib (400 mg daily) throughout the screening period.
* Clinically important intolerance or safety concerns with prior use of imatinib 400 mg daily.
* Prior treatment with an HSP90 inhibitor.
* Major surgery within 14 days prior to treatment with study drug, or failure to recover from the effects of such surgery.
* Wide field radiotherapy within 4 weeks prior to treatment with study drug, limited field radiation within 2 weeks, or failure to recover from such therapies.
* History of an ischaemic cardiac event or unstable cardiac disease within 3 months of study entry.
* QTc >450 ms using Fredericia's correction.
* Previous malignancy, except for basal cell and squamous cell skin carcinomas or carcinoma of the uterine cervix, unless treated with curative intent more than 2 years prior to study entry.
* Evidence of severe or uncontrolled systemic medical conditions which make it undesirable for the patient to take part in the study, or which could jeopardize protocol compliance. Patients with multiple comorbidities and/or requiring multiple concomitant medications (especially conditions/medications which may impair renal function or predispose to renal impairment) should be discussed with the Astex Medical Monitor at the discretion of the Investigator before enrollment.
* Prior history of infection with HIV, or known active hepatitis B or C viral infection (active screening for viral infections is not required for study entry).
* Significant visual impairment such that in the opinion of the investigator, further minor deterioration would have unacceptable consequences (eg. loss of ability to drive or live at home.
* The Safety Monitoring Committee may add other specific exclusion criteria to enhance the safety of the patients based on emerging safety data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-03; Primary Completion 2013-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Rate of reduction/stabilisation of tumour size at 4 months according to Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 criteria | 4 months

SECONDARY OUTCOMES:
Rate of reduction/stabilisation of tumour size at 6 months (6-month 'disease control rate' [DCR]), determined according to RECIST version 1.1 criteria. | 6 months
Progression-free survival at 6 months, and estimated proportion of patients surviving at 6 months. | 6 months
Objective responses, using RECIST version 1.1 criteria | 6 months
Changes in pharmacodynamic biomarkers assessed in tumour biopsies and plasma samples, and changes in tumour metabolism by Fludeoxyglucose - Positron emission tomography scans (FDG-PET). | 6 months
Relationships between KIT and PDGRFA tumour mutational status, changes in tumour dimensions, and exploratory pharmacodynamic biomarkers. | 6 months
Pharmacokinetic profile of AT13387 given in combination with imatinib. | 6 months
Treatment emergent adverse events, classified by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03. | 6 months

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Arizona Cancer Center at UMC North, Tucson, Arizona
  - Robert H. Lurie Cancer Center of Northwestern University, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health and Sciences University, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Wagner AJ, Agulnik M, Heinrich MC, Mahadevan D, Riedel RF, von Mehren M, Trent J, Demetri GD, Corless CL, Yule M, Lyons JF, Oganesian A, Keer H. Dose-escalation study of a second-generation non-ansamycin HSP90 inhibitor, onalespib (AT13387), in combination with imatinib in patients with metastatic gastrointestinal stromal tumour. Eur J Cancer. 2016 Jul;61:94-101. doi: 10.1016/j.ejca.2016.03.076. Epub 2016 May 5. PMID 27156227